CLINICAL TRIAL: NCT03426397
Title: Multicentre Evaluation of the "Wait-and-see" Policy for Complete Responders After Chemoradiotherapy for Rectal Cancer
Brief Title: "Wait-and-see" Policy for Complete Responders After Chemoradiotherapy for Rectal Cancer
Status: Recruiting | Type: Observational
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Dutch Cancer Society (Other)
Responsible Party: Sponsor
Other Study IDs: M16WAS
Record Dates: First submitted 2017-12-21; First posted 2018-02-08 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Rectal Neoplasms
Keywords: Complete response; Organ preservation; Wait-and-See; Watch-and-Wait; Watchful Waiting
MeSH Terms: conditions — Rectal Neoplasms; Pathologic Complete Response

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study population

SUMMARY:
The aim of this prospective observational cohort study is to provide short and long term oncological and functional outcome data on organ preserving treatment in good responders after a standard indication for neoadjuvant (chemo)radiation for rectal cancer.

DETAILED DESCRIPTION:
Standard treatment for patients with locally advanced rectal cancer consists of a long course of (CRT) followed by surgical resection. Although the aim of neoadjuvant treatment in these patients is not organ preservation, but rather to provide improved local control, in the tumour disappears completely. Studies from Maastricht, the UK and Brazil have shown that in selected patients with a clinical complete response after CRT, a "wait-and-see" policy without any surgery could be a safe alternative with comparable long-term outcome and better functional outcome compared to patients who had surgery.

The main objective of the study is to provide short and long term oncological and functional outcome data on organ preserving treatment in good responders after a standard indication for neoadjuvant (chemo)radiation. Additional aims are: to set up a national network with expertise centres in the 'wait-and-see' treatment of rectal cancer; to set up a national registry for organ preservation treatment that will generate more evidence on the management and oncological outcome of patients evaluated and treated with organ preservation and [3] to offer through this network to all patients who are considered good candidates this 'wait-and-see' approach using the most up to date tools for selection and follow-up.

Study design: multicenter prospective observational cohort study and implementation study. Study population: The population will consist of patients, aged 18 years or older, with rectal cancer who after a long course of CRT or a short course of radiation with a long waiting interval have a clinical complete response (ycT0N0).

The main study endpoint is 2-year non-regrowth disease-free survival. Secondary endpoints are [1] the number of fully operational centres who can deliver high quality organ preserving care in rectal cancer in the Netherlands, [2] 2-year regrowth rate, [3] 2-year local control, [4] 2-year overall survival, [5] determination of the optimal follow-up schedule and [6] quality of life.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: In the majority of patients who participate in the study, major surgery and the associated morbidity can be avoided. Although scientific proof shows "wait-and-see" only comes with a small risk with adequate selection and follow up, the exact risk is not yet well established and needs to be confirmed by this study. The benefit-risk ratio for this study is regarded as favourable.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Primary rectal cancer (pathologically confirmed)
* Treated with neoadjuvant (chemo)radiotherapy
* Clinical complete response (ycT0N0) to neoadjuvant treatment, as determined clinically (digital rectal examination, endoscopy) and radiologically (diffusion weighted imaging-MRI).
* Informed consent and capability of giving informed consent; before informed consent is obtained the patient will be extensively informed about the fact that 'wait-and-see' instead of conventional surgery is not accepted yet by most physicians and that the risks and benefits from these strategies have not been fully determined yet. These issues will be discussed in the patient information form as well.
* Comprehension of the alternative strategies and risks are clear to the patient (in other words that the patient understands the experimental base of the study).

Exclusion Criteria:

* Recurrent rectal cancer
* Contra-indications for MRI. If MRI is not possible because of contra-indications (e.g. pacemaker) patients will be excluded. MRI is crucial for response evaluation and follow-up and cannot be omitted in patients that follow the 'wait-and-see policy'.
* Unable to understand or read Dutch
* Unable or unwilling to comply to the intensive follow-up schedule

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population will consist of patients, aged 18 years or older, with rectal cancer who after a long course of CRT or a short course of radiation with a long waiting interval have a clinical complete response (ycT0N0), as determined by MRI (including DWI) and digital rectal examination + endoscopy. Only patients who fulfill the predefined list of criteria for a clinical complete response will be considered eligible for inclusion in the study.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2017-05-10 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
2-year non-regrowth disease-free survival | 2 years after start of wait-and-see protocol
  Absence of non-regrowth local or distant recurrence or death within 2 years of follow-up

SECONDARY OUTCOMES:
Number of fully operational centres | 2 years after start of wait-and-see protocol
  Number of operational centres who can deliver high quality organ preserving care in rectal cancer in the Netherlands
2-year local regrowth rate | 2 years after start of wait-and-see protocol
  The proportion of local regrowth
2-year local control | 2 years after start of wait-and-see protocol
  Absence of local recurrence(unresectable regrowth, resected with R1, or requiring more extensive than TME surgery) or death
2-year overall survival | 2 years after start of wait-and-see protocol
  Absence of death
Determination of the optimal follow-up schedule | 2 years after start of wait-and-see protocol
  A balance between early detection of recurrence and compliance to follow-up
Quality of life | At 3 months, 1 year, 2 years and 5 years after the start of wait-and-see protocol
  Quality of life (general health, disease specific and functional outcomes)

CONTACTS AND LOCATIONS:
Overall Officials: Geerard Beets, MD, PhD, Principal Investigator — Antoni van Leeuwenhoek - Netherlands Cancer Institute; Regina Beets -Tan, MD, PhD, Principal Investigator — Antoni van Leeuwenhoek - Netherlands Cancer Institute
Locations (14):
- Universitair Ziekenhuis Antwerpen, Antwerp, Belgium
- Netherlands (13):
  - Antoni van Leeuwenhoek, Amsterdam
  - VU Medisch Centrum, Amsterdam
  - Amphia Ziekenhuis, Breda
  - Deventer Ziekenhuis, Deventer
  - Westfriesgasthuis, Hoorn
  - Leeuwarden Medisch Centrum, Leeuwarden
  - Leiden University Medical Center, Leiden
  - Maastricht University Medical Centre, Maastricht
  - Radboud UMC, Nijmegen
  - Elisabeth Tweesteden Ziekenhuis, Tilburg
  - Diakonessenhuis, Utrecht
  - Universitair Medisch Centrum Utrecht, Utrecht
  - Isala Klinieken, Zwolle

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Meyer VM, Meuzelaar RR, Schoenaker IJH, de Groot JB, Reerink O, de Vos Tot Nederveen Cappel WH, Beets GL, van Westreenen HL. Delayed TME Surgery in a Watch-and-Wait Strategy After Neoadjuvant Chemoradiotherapy for Rectal Cancer: An Analysis of Hospital Costs and Surgical and Oncological Outcomes. Dis Colon Rectum. 2023 May 1;66(5):671-680. doi: 10.1097/DCR.0000000000002259. Epub 2021 Nov 24. PMID 34856587